CLINICAL TRIAL: NCT03488745
Title: Examining an App-based Mental Health Intervention for Cancer Patients and Caregivers
Brief Title: Addressing Mental Health of Cancer Patients and Caregivers Using a Mobile App Suite
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Philip Chow, Ph.D., Assistant Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20403
Record Dates: First submitted 2018-03-20; First posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Mental Health Wellness 1; Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IntelliCare + Phone Coaching (Experimental): Participants will receive IntelliCare apps with phone coaching for 7 weeks. In this arm, participants will pick two IntelliCare apps to use every week. Participants will receive a phone coaching call before they use the apps, for approximately 30 minutes, as well as 3 weeks after initiating app use (10 minute call).
  Interventions: Behavioral: IntelliCare + Phone Coaching

INTERVENTIONS:
Behavioral: IntelliCare + Phone Coaching — IntelliCare is composed of 13 separate, native apps. Each app targets a specific aspect of mental health (e.g., reducing worry, increasing social support, tracking negative thoughts). The apps are available to the public in both Android and iPhone stores. Participants will be asked to try two new IntelliCare apps every week, for 7 weeks. Phone coaching will occur at Day 0, before using any of the apps, and the third week of app usage.

SUMMARY:
A cancer diagnosis affects not only patients but also their caregivers. The purpose of this study is to test the feasibility of using a mobile app suite, IntelliCare, to improve the mental health of cancer patients and caregivers.

DETAILED DESCRIPTION:
Cancer patients and/or their caregivers will receive access to the mobile app suite, IntelliCare, as well as phone coaching that will focus on how to use the apps. IntlliCare is composed of separate apps that each target a specific aspect of mental health (e.g., reducing worry). The apps are interactive and designed for users to engage in short time bursts (e.g., less than a minute). IntelliCare was originally designed to be paired with phone coaching that focuses on how to use the apps and overcome barriers to usage.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to comply with scheduled visits and study procedures.
* Caregiver/support person of patient undergoing treatment for cancer in the Breast Care Clinic OR patient undergoing treatment for cancer in the Breast Care Clinic
* Owns a smart phone or they are willing to carry one during the study if one is provided.

Exclusion Criteria:

* Under 18 years old
* Non-English Speaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-03-27 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Depression Symptoms | Change in depression symptoms from baseline to post-intervention (7 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System 4-Item Depression Scale (from 29-item Profile), measures depression on a continuous scale. Scores on this scale range from 4-20, with a higher score indicating greater severity of depression.
Anxiety Symptoms | Change in anxiety symptoms from baseline to post-intervention (7 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System 4-Item Anxiety Scale (from 29-item Profile), measures anxiety on a continuous scale. Scores on this scale range from 4-20, with a higher score indicating greater severity of anxiety.
Clinical Mood Symptoms | Change in clinical mood symptoms from baseline to post-intervention (7 weeks after baseline)
  Patient Health Questionnaire-4 contains measures clinical symptoms of mood and anxiety disorders. Scores on this scale range from 0-12, with a higher score indicating greater severity of mood symptoms. Unlike the Patient-Reported Outcomes Measurement Information System scales, this scale has pre-determined clinical cutoffs for mild, moderate, and severe symptoms, which will be used to classify severity of mood symptoms.

SECONDARY OUTCOMES:
Physical Function | Change in physical function from baseline to post-intervention (7 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System 4-Item Physical Function Scale (from 29-item Profile). Scores on this scale range from 4-20, with a higher score indicating less impairment of physical function.
Life Meaning/purpose | Change in life meaning/purpose from baseline to post-intervention (7 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System 4-Item Life Meaning and Purpose Scale. Scores on this scale range from 4-20, with a higher score indicating more life meaning and purpose.
Sleep Quality | Change in sleep disturbance from baseline to post-intervention (7 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System 4-Item Sleep Disturbance Scale (from 29-item Profile). Scores on this scale range from 4-20, with a higher score indicating more sleep disturbance.
Fatigue | Change in fatigue from baseline to post-intervention (7 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System 4-Item Fatigue Scale (from 29-item Profile). Scores on this scale range from 4-20, with a higher score indicating more fatigue.
Pain Interference | Change in Pain Interference from baseline to post-intervention (7 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System 4-Item Fatigue Scale (from 29-item Profile). Scores on this scale range from 4-20, with a higher score indicating more pain interference in daily life.
Patient Health Care Utilization | Change in Patient Health Care Utilization from baseline to post-intervention (7 weeks after baseline)
  Created a scale since none currently exist. Items (in order) are the following:
  1. Over the past two months, how many times did you go to the emergency department?
  2. Were any of these visits related to your side effects from cancer treatment? (Yes/No/I Don't Know)
  3. How many visits were related to side effects from cancer treatment?
  4. Over the past two months, did you ever miss a scheduled appointment for cancer treatment? (Yes/No/I Don't Know)
  5. How many appointments did you miss?
  6. Over the past two months, have you used any cancer support services? These include programs for emotional support, or services for transportation, lodging, or other needs related to cancer treatment. (Yes/No/I Don't Know)
  7. What types of services have you used?
Caregiver Health Care Utilization | Change in Caregiver Health Care Utilization from baseline to post-intervention (7 weeks after baseline)
  Created a scale since none currently exist. Items (in order) are the following:
  1. Over the past two months, how many times did you go to the emergency department?
  2. Over the past two months, how many times did you visit your primary care doctor for anything OTHER THAN routine care?
  3. Over the past two months, have you used any cancer support services? These include programs for emotional support, or services for transportation, lodging, or other needs related to caregiving for your loved one with cancer. (Yes/No/I Don't Know)
  4. What types of services have you used?
Ability to Participate in Social Roles and Activities | Change in Ability to Participate in Social Roles and Activities from baseline to post-intervention (7 weeks after baseline)
  Patient-Reported Outcomes Measurement Information System 4-Item Ability to Participate in Social Roles and Activities Scale (from 29-item Profile). Scores on this scale range from 4-20, with a higher score indicating more ability to participate in social roles and activities in daily life.
Caregiver Self-Efficacy | Change in Caregiver Self-Efficacy from baseline to post-intervention (7 weeks after baseline)
  Caregiver Self-Efficacy Scale (CaSES; Ugalde, Krishnasamy, & Schofield, 2013). A 21-item scale developed to measure self-efficacy in informal cancer caregivers. Scores range from 0-84, with a higher score indicating more self-efficacy.

OTHER OUTCOMES:
Positive and Negative Mood | Surveys administered during the following weeks: 1, 2, 3, 4, 5, 6, 7
  Overall, how have you felt over the past week? (Scale from 1=Very negative to 5=Very positive)
Drug Use | Surveys administered during the following weeks: 1, 2, 3, 4, 5, 6, 7
  How much have you used alcohol or tobacco to cope with negative feelings? (Scale from 1=Not at all to 5=A lot or extremely)
Pain | Surveys administered during the following weeks: 1, 2, 3, 4, 5, 6, 7
  How much physical pain have you experienced? (Scale from 1=Not at all to 5=A lot or extremely)
Social Connectedness | Surveys administered during the following weeks: 1, 2, 3, 4, 5, 6, 7
  1. How connected did you feel to family and friends? (Scale from 1=Not at all to 5=A lot or extremely)
  2. How much support did you receive from loved ones? (Scale from 1=Not at all to 5=A lot or extremely)
  3. How much were you able to support loved ones? (Scale from 1=Not at all to 5=A lot or extremely)
Anhedonia | Surveys administered during the following weeks: 1, 2, 3, 4, 5, 6, 7
  How much interest or pleasure did you have in doing things? (Scale from 1=Not at all to 5=A lot or extremely)
Anxiety | Surveys administered during the following weeks: 1, 2, 3, 4, 5, 6, 7
  How much did you feel nervous, anxious, or on edge? (Scale from 1=Not at all to 5=A lot or extremely)
Physical Activity | Surveys administered during the following weeks: 1, 2, 3, 4, 5, 6, 7
  How active were you? (Scale from 1=Not at all to 5=A lot or extremely)
Emotion Regulation | Surveys administered during the following weeks: 1, 2, 3, 4, 5, 6, 7
  How well have you managed negative feelings? (Scale from 1=Not at all to 5=A lot or extremely)
Future Positive and Negative Mood | Surveys administered during the following weeks: 1, 2, 3, 4, 5, 6, 7
  Overall, how do you expect to feel next week? (Scale from 1=Very negative to 5=Very positive)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Chow, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chow PI, Showalter SL, Gerber MS, Kennedy E, Brenin DR, Schroen AT, Mohr DC, Lattie EG, Cohn WF. Use of Mental Health Apps by Breast Cancer Patients and Their Caregivers in the United States: Protocol for a Pilot Pre-Post Study. JMIR Res Protoc. 2019 Jan 14;8(1):e11452. doi: 10.2196/11452. PMID 31344674